CLINICAL TRIAL: NCT01948843
Title: Phase 1 Trial of ADI-PEG 20 Plus Doxorubicin in Patients With HER2 Negative Metastatic Breast Cancer or Advanced Solid Tumor
Brief Title: Ph 1 ADI-PEG 20 Plus Doxorubicin; Patients With HER2 Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLARIS2013-004
Record Dates: First submitted 2013-09-11; First posted 2013-09-24 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: HER2 Negative Metastatic Breast Cancer
Keywords: HER2 Negative Metastatic Breast Cancer
MeSH Terms: interventions — ADI PEG20

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADI-PEG 20 (Experimental): arginine deiminase formulated with polyethylene glycol
  Interventions: Drug: ADI-PEG 20

INTERVENTIONS:
Drug: ADI-PEG 20

SUMMARY:
Certain cancers require the amino acid arginine. Arginine deiminase (ADI) is an enzyme from microbes that degrade arginine. ADI has been formulated with polyethylene glycol, and has been used to treat patients that have cancers that require arginine. In this study, ADI will be combined with the well known chemotherapy Doxorubicin and the safety and potential efficacy of this combination will be explored in patients with HER2 Negative Metastatic Breast Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven HER2 negative metastatic breast cancer (dose escalation portion and MTD expansion portion) or advanced solid tumor (dose escalation portion).
2. ASS deficiency (defined as <50% ASS expression) demonstrated on tissue specimen by Immunohistochemistry (IHC). Cytology and fine need aspirate specimens are not acceptable for ASS testing.
3. Unresectable disease or subject refused surgery.
4. Measurable disease as assessed by RECIST 1.1 criteria (Appendix A).
5. Failed available therapy known to confer clinical benefit but no more than 4 prior lines of chemotherapy for metastatic disease.
6. Time to treatment failure from doxorubicin containing regimen ≥ 12 months if previously treated with doxorubicin.
7. Age ≥ 18 years.
8. ECOG performance status of 0 - 2. -

Exclusion Criteria:

1. Serious infection requiring treatment with systemically administered antibiotics at the time of study entrance, or an infection requiring systemic antibiotic therapy within 7 days prior to the first dose of study treatment.
2. Prior epirubicin exposure of > 600 mg/m2.
3. Pregnancy or lactation.
4. Expected non-compliance.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV), cardiac arrhythmia, or psychiatric illness, social situations that would limit compliance with study requirements.
6. Subjects who have had any anticancer treatment prior to entering the study and have not recovered to baseline (except alopecia) or ≤ Grade 1 AEs, or deemed irreversible from the effects of prior cancer therapy. AEs > Grade 1 that are not considered a safety risk by the Sponsor and Investigator may be allowed upon agreement with both.
7. Subjects with history of another primary cancer, including co-existent second malignancy, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present in the opinion of the Investigator will not affect subject outcome in the setting of breast cancer diagnosis.
8. Subjects who had been treated with ADI-PEG 20 previously.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 2 years estimated - course of study
  Assessment of safety and tolerability of ADI-PEG 20 in combination with doxorubicin in HER2 negative metastatic breast cancer
Determine preliminary estimates of efficacy, measured by RECIST 1.1 criteria, for ADI-PEG 20 combo with doxorubicin in HER2 negative metastatic breast cancer. | 2 years estimated - course of study

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, MD, Principal Investigator — MD Anderson
Locations (1):
- M.D. Anderson Cancer Center, Houston, Texas, United States